CLINICAL TRIAL: NCT04870385
Title: An Islamic Psychospiritual-Acceptance and Commitment-based Prevention Program for At-Risk Young Adults in the COVID-19 Pandemic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: International Islamic University Malaysia (Other)
Collaborators: International Institute of Islamic Thought (Unknown)
Responsible Party: Principal Investigator, Jamilah Hanum Abdul Khaiyom, PhD, Assistant Professor, International Islamic University Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SPI21-052-0052
Record Dates: First submitted 2021-04-07; First posted 2021-05-03 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Psychological Distress
Keywords: Acceptance and Commitment Therapy (ACT); Islamic psychospiritual intervention; Online intervention; COVID-19; Prevention program
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: A randomised parallel interventional study model in which there will be 2 groups, an intervention group and a waitlist control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): 5-week online prevention program
  Interventions: Behavioral: 5-week prevention program
- Control (Other): Waitlist control
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: 5-week prevention program — Online modular psychological prevention program featuring integrated elements of Islamic spirituality and Acceptance and Commitment Therapy (ACT).
  Arms: Treatment
Behavioral: Control — Control group waitlisted to receive prevention program after completion of final data collection.
  Arms: Control

SUMMARY:
The COVID-19 pandemic has increased mental health concerns worldwide, and young adults are at higher risk of experiencing increased psychological distress due to the pandemic. University students face compounding stressors during the pandemic, such as online and remote learning, economic insecurity, and uncertain career prospects. This study aims to evaluate the effectiveness of an online modular prevention program featuring integrated elements of Acceptance and Commitment Therapy (ACT) and Islamic spirituality in reducing the psychological distress and increasing the psychological flexibility, self-compassion, and resilience of Muslim university students in Malaysia.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate or postgraduate student enrolled in a Malaysian university
* aged 18-29 years old
* Obtained moderate and above levels in either one of the stress, anxiety, and depression subscales of the DASS-21 pre-intervention assessment
* Muslim
* Owns a gadget with Internet access
* Can read and understand English

Exclusion Criteria:

* Those with previous experience with a modular ACT-based treatment with Islamic elements
* Those with past or present diagnosis of mental/neurological disorder
* Those reporting active suicidality
* Those involved in any other form of psychological treatment (ie. psychotherapy, pharmacotherapy)

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-04-11 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Changes in psychological distress | Measured at pre-intervention, mid-intervention (third week of prevention program), post-intervention (up to 1-week after completion of program), and 1-month follow-up
  Measured using the Depression, Anxiety, and Stress Scale (DASS-21; Lovibond & Lovibond, 1995).

SECONDARY OUTCOMES:
Changes in psychological flexibility | Measured at pre-intervention, mid-intervention (third week of prevention program), post-intervention (up to 1-week after completion of program), and 1-month follow-up
  Measured using the Acceptance and Action Questionnaire (AAQ-II; Bond et al., 2011; Hayes et al., 2004).
Changes in self-compassion. | Measured at pre-intervention, mid-intervention (third week of prevention program), post-intervention (up to 1-week after completion of program), and 1-month follow-up
  Measured through the Self-Compassion Scale (SCS; Neff 2003; Neff, 2015).
Changes in resilience | Measured at pre-intervention, mid-intervention (third week of prevention program), post-intervention (up to 1-week after completion of program), and 1-month follow-up
  Measured by the Brief Resilience Scale (BRS; Smith et al., 2008).

CONTACTS AND LOCATIONS:
Overall Officials: Jamilah Hanum Abdul Khaiyom, PhD, Principal Investigator — International Islamic University Malaysia
Locations (1):
- International Islamic University Malaysia, Kuala Lumpur, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No